CLINICAL TRIAL: NCT05846971
Title: Clinical Utility of Methylation-based Prognostic Assay for Barrett's Esophagus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Capsulomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 23-001
Record Dates: First submitted 2022-11-14; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Barrett Esophagus; Esophageal Cancer
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group will receive standard-of-care clinical data for their virtual patient cases. No educational material on the methylation assay will be provided.
- Intervention Group (Experimental): The intervention group will receive standard-of-care clinical data for their virtual cases along with educational materials about the methylation assay. This group will then be provided with methylation assay data to be used in addition to clinical data.
  Interventions: Other: Educational materials on validated methylation assay

INTERVENTIONS:
Other: Educational materials on validated methylation assay — Educational materials include overall information on the assay including what the test does, how to use the test and report, and performance metrics on the test.
  Arms: Intervention Group

SUMMARY:
Capsulomics has developed a prognostic assay for patients with diagnosed Barrett's esophagus (BE). This study will measure how gastroenterologists make surveillance and treatment management decisions when presented with different clinical and prognostic assay information.

DETAILED DESCRIPTION:
Capsulomics has developed a prognostic assay for patients with diagnosed Barrett's esophagus (BE). This study will measure how gastroenterologists make surveillance and treatment management decisions for virtual patient cases when presented with different clinical and prognostic assay information. The data from this study will be published in a peer-review scientific journal.

ELIGIBILITY:
Inclusion Criteria:

1. Be currently practicing board-certified gastroenterologist practicing in the United States
2. Have practiced (as a board-certified gastroenterologist) for greater than 2
3. Be English-speaking
4. Have ≥ 50 Barrett's esophagus patients under care annually
5. Have Internet access
6. Have no prior experience with the methylation assay test
7. Provide voluntary informed consent to participate in the study.

Exclusion Criteria:

1. Non-practicing gastroenterologists
2. Less than two years of gastroenterology practice
3. Non-English speaking
4. Does not have access to the internet
5. Does not consent to participate in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical performance change in physician behavior. | 1 year
  Change in the overall and the diagnostic and treatment in patient simulations: difference-in-differences regression analysis between the control and the intervention groups' diagnosis and treatment of risk progression in patients with Barrett's esophagus, as measured by the participants' diagnostic and treatment scores. In each category, participants' care recommendations are evaluated, ranging from 0 to a high potential score of up to 10, where higher scores mean increased intensity in surveillance and treatment, to measure the impact of the methylation assay on care decision making.
The impact of methylation assay on physician confidence in clinical care decision-making. | 1 year
  Measure the confidence in care decisions based on patient's methylation test result: Once the intervention group is exposed to the intervention, education materials on the methylation assay (a validated molecular test for risk stratifying patients with Barrett's esophagus), the scores are measured, on a scale of 0 to 10 from round 1 (pre-exposure) to round 2 (post-exposure) and observe how the assay impacts confidence in the physician following evidence-based patient care.

CONTACTS AND LOCATIONS:
Locations (1):
- Capsulomics, Inc., Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No